CLINICAL TRIAL: NCT00364598
Title: A Phase I Open Label Pilot Study to Obtain Tissue for Histological Analysis After Application of Anginera™ in Adults With A Left Ventricular Assist Device As A Bridge To Transplant
Brief Title: Study of Anginera in Adults With a Left Ventricular Assist Device (LVAD) as Bridge to Transplant
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theregen, Inc. (Industry)
Responsible Party: Gary Gentzkow, M.D. Chief Medical Officer, Theregen, Inc.
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TI-102
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Heart Failure
Keywords: Anginera; LVAD; Transplant; Histology; LVAD implantation as a bridge to transplant
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anginera, a human tissue replacement therapy

SUMMARY:
The purpose of this study is to obtain human heart tissue after treatment with Anginera to determine its effect on a variety of things that might indicate improvement in heart function. Patients who will have a left ventricular assist device (LVAD) implanted while they wait for a donated heart will be treated with Anginera. At the time of heart transplant, their diseased heart which is removed will be analyzed by microscopic examination to see what effect Anginera had.

DETAILED DESCRIPTION:
This will be a prospective, multi-center, randomized, open-label, within-patient paired design study. The primary purpose is to analyze cardiac tissue obtained after application of Anginera to adults with an LVAD as a bridge to transplant, to determine effects on various markers.

ELIGIBILITY:
Inclusion Criteria:

* Stage D Heart Failure
* Patients having an LVAD implanted as a bridge to transplant.

Exclusion Criteria:

* Biopsy proven acute myocarditis
* Known Giant Cell Myocarditis
* Known infiltrative disease, e.g. cardiac Amyloidosis, Sarcoidosis, hemochromatosis, Fabry's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
To analyze cardiac tissue obtained after application of Anginera to adults with an LVAD as a bridge to transplant, to determine effects on various markers.

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth B Margulies, M.D., Principal Investigator — University of Pennsylvania; Y. Joseph Woo, M.D., Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania